CLINICAL TRIAL: NCT00326482
Title: A Pilot Study of Hepatic Fibrosis in HIV/AIDS Patients With Chronically Elevated Transaminases on Antiretroviral Therapy
Brief Title: Liver Fibrosis in HIV-Infected Patients With Elevated Liver Enzymes on Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060153; 06-I-0153
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01-06

CONDITIONS: Liver Fibrosis; Steatohepatitis; Elevated Transaminases
Keywords: Drug Toxicity; Steatohepatitis; Hepatotoxicity; Liver Biopsy; Liver Disease; Natural History; HIV; Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Drug-Related Side Effects and Adverse Reactions; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prior Liver Biopsy: HIV+ historical liver biopsy history
- Prospective Liver Biopsy with ARV: HIV+ taking c/ARV medications
- Prospective Liver Biopsy without ARV: HIV+ not taking c/ARV medications

SUMMARY:
This study will provide a basis for research on the impact of liver injury caused by antiretroviral therapy in HIV-infected patients. Elevated liver enzymes called AST and ALT are common in HIV-infected patients taking antiretroviral medications and can indicate liver damage. Although there are a number of possible causes for these elevations, such as infections with a hepatitis virus, antiretroviral medications alone can lead to the elevations. The study will focus particularly on evidence of liver fibrosis, which is a sign of progressive liver damage.

HIV-infected patients 18 and older who 1) have been taking combination antiretroviral therapy for at least 12 months and have been on a stable regimen for at least 3 months, and 2) have had elevated AST or ALT levels for at least 6 months may be eligible for this study. Patients who have had liver biopsies performed in the past may be eligible for participation.

Participants undergo the following tests and procedures over a 12-month period:

* Oral glucose tolerance test: The patient drinks a glucose (sugar) drink. Blood samples are then drawn over 2 hours through an intravenous (IV) line in the patient's arm. This test measures how high the patient's blood sugar and insulin levels rise after drinking a standard glucose load.
* Transient elastography: This ultrasound test uses vibration (sound waves) to measure liver stiffness (fibrosis). Vibrations move faster through a fibrotic liver.
* Triple-phase CT scan and single slice CT scan of L4-5: Patients fast for 4 hours before the CT scan. A contrast material is injected through a catheter placed in an arm vein to improve the visibility of the liver in the specialized X-ray images obtained in the CT scanner.
* Liver biopsy: This test removes a small sample of liver tissue for microscopic examination, particularly for evidence of fibrosis. The skin over the biopsy site is numbed and a needle is passed through the skin and rapidly in and out of the liver. Patients may be given a sedative for the procedure.
* Follow-up visits. Patients return for follow-up visits 1 to 4 weeks after the liver biopsy and three more times over the course of the study for a medical history, physical examination and blood tests.

Patients may participate in an additional 4-year follow-up, during which they have visits every 3-12 months and are offered the opportunity to repeat the biopsy no sooner than 1 year after the first biopsy.

DETAILED DESCRIPTION:
At present, there are no clear guidelines as to when antiretroviral therapy for human immunodeficiency virus (HIV) infection should be stopped in the setting of elevated liver enzymes. In large part, this is due to a limited understanding of the natural history of antiretroviral-related hepatotoxicity. Although several antiretrovirals have been reported to cause fatal acute hepatitis, more often they cause an asymptomatic elevation in transaminase levels, the optimal management of which is uncertain. This pilot study seeks to create a foundation for research on the impact of antiretroviral-induced liver injury by providing an estimate of the prevalence of hepatic fibrosis in a cohort of sixty HIV-infected patients who have chronically elevated transaminases while on antiretroviral therapy in the absence of chronic hepatitis B (HBV) or C (HCV) coinfection. Liver biopsy specimens will be evaluated for fibrosis by microscopic examination, the current gold standard for assessing the nature and severity of liver disease.[1] The presence of fibrosis, as well as other histopathology, will be described using a validated scoring system. Primarily, this will be a crosssectional study, but subjects will be offered the opportunity to participate in an extended follow-up period and undergo another liver biopsy. Individuals will not be excluded on the basis of alcohol abuse, insulin resistance, or lipodystrophy, but data will be collected on these potentially confounding variables. Noninvasive measures, such as transient elastography (an ultrasonic technique), will be assessed for their ability to predict fibrosis in this population. Correlations will also be sought with laboratory markers of fibrosis. The identification of fibrosis (and its precursors) in association with antiretroviral therapy may be very clinically relevant as it may slowly regress with cessation of the causal agent(s). If the causal agent is continued, however, cirrhosis may develop, the reversal of which is thought to be rare.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 years or older.

Ability to understand and willingness to provide written informed consent.

Willingness to undergo liver biopsy.

Willingness to comply with study requirements and procedures including storage of blood and liver tissue samples for use in future studies of HIV, AIDS, immune function, hepatic diseases, or other related diseases.

Established HIV diagnosis (documentation of HIV-1 infection by licensed ELISA testing and confirmed by Western Blot).

For the antiretroviral cohort on combination antiretroviral therapy for at least 12 months with stable regimen for at least 3 months prior to enrollment.

Chronically elevated transaminases for at least 6 months documented by an elevated AST and/or ALT on the following 3 occasions within the 12 months prior to enrollment:

1. Screening;
2. Less than 6 months (24 weeks) prior to enrollment (distinct from screening);
3. More than 6 months prior to enrollment.

   Note: Occasions must be at least 8 weeks apart.

   Specific screening lab criteria:
   * AST and/or ALT greater than upper limit of normal;
   * Absolute neutrophil count greater than 750/mm(3);
   * PT/PTT within normal range;
   * Platelets greater than 50,000/uL;
   * Hemoglobin greater than or equal to 10 mg/dL;
   * Creatinine less than or equal to 2.0 mg/dL;
   * Negative serum or urine pregnancy test for females of childbearing potential.

   Willingness to avoid medications that contain aspirin for 7 days PRIOR to liver biopsy and nonsteroidal anti-inflammatory drugs for 3 days PRIOR to liver biopsy.

   Willingness to avoid medications that contain aspirin for a week AFTER liver biopsy.

   Willingness to avoid other medications or herbal supplements (e.g., gingko biloba) which may increase the risk of bleeding before and after liver biopsy, as directed by the study team.

   Willingness to restrict activity for 72 hours after liver biopsy.

   Have a primary care physician.

   HIV monoinfected individuals who have had a previous liver biopsy to evaluate chronically elevated transaminases on antiretroviral therapy or for another indication may be allowed to enroll in the study for the purposes of obtaining additional information on predictors of liver disease and to observe the natural history. In such instances, investigators will attempt to access this tissue for review.

   EXCLUSION CRITERIA:

   Chronic hepatitis B infection (defined as positive HBsAg or hepatitis B viral load greater than 10,000 copies/ml).

   Hepatitis C infection (defined as positive HCV viral load) or history of treatment for chronic hepatitis C.

   Acute Hepatitis A infection (defined as HAV IgM positive).

   Suspected rhabdomyolysis (e.g., markedly elevated AST with elevated CPK).

   Known or suspected autoimmune hepatitis.

   Known or suspected biliary diseases, such as primary biliary cirrhosis or sclerosing cholangitis.

   Known or suspected Wilson's disease, alpha-1-antitrypsin deficiency, celiac disease.

   History of primary hemochromatosis, glycogen storage disease, amyloidosis, or cystic fibrosis.

   Clinical evidence of decompensated liver disease (e.g., jaundice, ascites, esophageal varices, or hepatic encephalopathy).

   Active clinical pancreatitis.

   Chronic renal disease.

   Morbid obesity (BMI greater than or equal to 40), if judged to be a contradiction to percutaneous liver biopsy

   AFP greater than or equal to 100 ng/mL.

   Hepatoma or hepatocellular carcinoma.

   Pregnancy.

   Active opportunistic infection (except oral thrush) or neoplasm (except Kaposi's sarcoma, skin cancer, or cancer of the cervix or anus, unless known or suspected liver metastasis).

   Severe psychiatric disorder that would interfere with adherence to protocol requirements. Individuals who have a stable psychiatric condition may be eligible.

   Decompensated cardiac or pulmonary disease limiting physical activity (e.g., New York Heart Association Heart Failure Class 2 or higher).

   History of unexplained bleeding.

   Allergy to lidocaine.

   Current use or a history of treatment with interleukin-2, interferon-alpha or other investigational agent(s) within 6 months of protocol screening. However, antiretroviral medication obtained through expanded access programs are permitted.

   Current use or a history of treatment with a systemic corticosteroid, immunosuppressive or cytotoxic agent within 90 days of protocol screening. However, volunteers receiving no more than one day of corticosteroid therapy in the 90 days prior to screening will be eligible.

   Any medical condition for which an investigator believes liver biopsy may be contraindicated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients with chronically elevated transaminases while on c/ARV medications or not on c /ARV medications that agree to research procedures that investigate the prevalence of hepatic fibrosis in the absence of hepatitis B or C co-infection@@@
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2006-07-31 (Actual)

PRIMARY OUTCOMES:
Presence of hepatic fibrosis on liver biopsy as measured histologically by stage | At study entry, potential for repeat liver biopsy staging during longitudinal follow-up
  Liver Biopsy Scoring

SECONDARY OUTCOMES:
Liver biopsy evidence of hepatic steatosis as measured by degree (0 to 4), character and location | At study entry, potential for repeat liver biopsy staging during longitudinal follow-up
  Liver Biopsy Scoring
Liver biopsy evidence of hepatic inflammation by type and severity | At study entry, potential for repeat liver biopsy staging during longitudinal follow-up
  Liver Biopsy Scoring
Correlation between histopathologic findings on liver biopsy and clinical, laboratory and radiologic parameters | At study entry, longitudinally
  Liver Biopsy Scoring

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sulkowski MS, Thomas DL, Chaisson RE, Moore RD. Hepatotoxicity associated with antiretroviral therapy in adults infected with human immunodeficiency virus and the role of hepatitis C or B virus infection. JAMA. 2000 Jan 5;283(1):74-80. doi: 10.1001/jama.283.1.74. PMID 10632283
- [Background] Crum-Cianflone N, Collins G, Medina S, Asher D, Campin R, Bavaro M, Hale B, Hames C. Prevalence and factors associated with liver test abnormalities among human immunodeficiency virus-infected persons. Clin Gastroenterol Hepatol. 2010 Feb;8(2):183-91. doi: 10.1016/j.cgh.2009.09.025. Epub 2009 Oct 2. PMID 19800985
- [Background] Ingiliz P, Valantin MA, Duvivier C, Medja F, Dominguez S, Charlotte F, Tubiana R, Poynard T, Katlama C, Lombes A, Benhamou Y. Liver damage underlying unexplained transaminase elevation in human immunodeficiency virus-1 mono-infected patients on antiretroviral therapy. Hepatology. 2009 Feb;49(2):436-42. doi: 10.1002/hep.22665. PMID 19085967
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-I-0153.html